CLINICAL TRIAL: NCT00158015
Title: Prospective Minnesota Study of ECHO Tissue Doppler Imaging in Cardiac Resynchronization Therapy
Status: Completed | Type: Observational
Sponsor: Hennepin Healthcare Research Institute (Other)
Collaborators: Guidant Corporation (Industry)
Responsible Party: Steven R. Goldsmith, Minneapolis medical research foundation
Other Study IDs: 1886-4
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2012-10-04 (Estimated); Status verified 2012-10

CONDITIONS: Heart Failure
Keywords: Echocardiography; tissue Doppler Imaging; Cardiac Resynchronization Therapy
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to assess whether tissue doppler imaging is useful in predicting which patients will respond most to Cardiac Resynchronization therapy ( a type of pacemaker)

DETAILED DESCRIPTION:
Cardiac Resynchronization Therapy (CRT) is a newly developed therapy designed to improve outcomes in patients with heart failure(HF). Recent studies have shown significant symptomatic improvement and a decrease in hospitalization and mortality with CRT. However, up to 30 % of patients do not experience improvement with this invasive and costly therapy. Tissue Doppler Imaging (TDI) is emerging as an effective tool for non-invasively assessing mechanical dyssynchrony of the left ventricle (LV) and may aid in the identification of LV mechanical dyssynchrony to predict clinical response to CRT. PROMISE-CRT is designed to address the following hypothesis: Changes in tissue doppler imaging measures of left ventricular mechanical dyssynchrony from baseline to one week following cardiac resynchronization therapy will correlate with the clinical response at three months. Seventy HF patients clinically indicated to receive CRT will be enrolled in this six-month multi-center study conducted in the Minneapolis-St. Paul metropolitan area. TDI analyses, measures of clinical improvement and LV remodeling will be conducted one week, three months, six months after CRT implementation.

ELIGIBILITY:
Inclusion Criteria:

Moderate or severe heart failure defined as NYHA class III-IV despite optimal pharmacological heart failure therapy.

Stable Heart failure as defined as not hospitalized within the last month. A 12 lead electrocardiogram (ECG) obtained no more than 90 days prior to enrollment documenting a sinus rate >50bpm, QRS duration >120ms and PR interval> 150ms Ejection Fraction <35% documented within the last 6 months by one of the following methods: echo ( standard or TEE) LV gram, or MUGA Clinically indicated to receive CRT Ability to complete all the study visits including geographic stability

Exclusion criteria:

Serum creatinine >3.5 Have or had a Myocardial infarct, unstable angina, percutaneous coronary intervention or coronary artery bypass graft during the preceding 30 days prior to enrollment.

Have had previous cardiac resynchronization therapy, a coronary venous pace/sense lead or attempted LV lead placement.

Dyspnea believed by the physician to be primarily related to lung disease. Have an atrial tachyarrhythmia that is permanent ( ie does not terminate spontaneously and cannot be terminated with medical intervention)or persistent (can be terminated with medical intervention but does not terminate spontaneously)within 90 days prior to enrollment Poor sinus node function that MD predicts will require >70% atrial pacing. Inability to perform the six minute walk. Life expectancy of less than 6 months due to other medical conditions or expected to undergo heart transplant within the next 6 months.

Have a mechanical tricuspid heart valve. Hypertrophic obstructive cardiomyopathy. Patients with a hypersensitivity to a 0.7mg nominal dose of dexamethasone. Surgically uncorrected primary valvular heart disease. Patients who are currently enrolled in another investigational study that would directly impact the treatment or outcome of the current study.

Patients who are younger than 18 years of age, pregnant, or who are mentally incompetent and cannot sign a patient informed consent.

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stable Heart failure subjects receiving CRT
Sampling Method: Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2004-10; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan J Bank, MD, Principal Investigator — St. Paul Heart Clinic
Locations (7):
- United States (7):
  - Metropolitan Cardiology consultants, Coon Rapids, Minnesota
  - Minnesota Heart Clinic, Edina, Minnesota
  - Minneapolis Heart Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - St. Paul Heart Clinic, Saint Paul, Minnesota
  - University of Wisconsin, Madison, Wisconsin